CLINICAL TRIAL: NCT00214162
Title: Web-based Support for Informal Caregivers in Cancer
Brief Title: CHESS Caregivers Study: Web-based Support for Informal Caregivers in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2002-436; 1R01NR008260-01 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer; Prostate Cancer
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): internet access and computer for 1 year
  Interventions: Behavioral: computer with internet
- 2 (Experimental): computer and Full CHESS
  Interventions: Behavioral: Comprehensive Health Enhancement Support System

INTERVENTIONS:
Behavioral: Comprehensive Health Enhancement Support System — Full CHESS
  Arms: 2
Behavioral: computer with internet — computer with internet use x 1 year
  Arms: 1

SUMMARY:
Web-Based Support for Informal Caregivers in Cancer Brief Summary (including hypothesis):

Informal caregivers need information, skills and emotional support to address physical, spiritual, and emotional needs associated with chronic illnesses including late stage cancer. Unfortunately, current conditions force clinicians to reduce their interaction time with patients and informal caregivers. Complimentary methods must be developed to provide needed information and support to caregivers. The proposed research will measure and explain the impact of two computer-based support systems that meet caregiver needs and facilitate information exchange with clinicians. The system, CHESS (Comprehensive Health Enhancement Support System) is a non-commercial computer system that provides patients with disease specific information, emotional support and skill building tools. In the expanded form to be tested in this study, CHESS with Caregiver Support (CGCHESS) will also provide the caregiver with more information, support and skills training related to palliative care. CGCHESS will be further enhanced to communicate essential patient and caregiver information to clinicians prior to a scheduled clinic visit and when patient symptoms exceed a threshold.

The investigators' primary hypothesis is that CGCHESS + Clinician Report (CR) will reduce caregiver burden more than CGCHESS because of the additional support caregivers and patients receive from clinicians who have access to the CHESS clinician report. Secondary analyses will study the mechanisms of the CHESS effect. Specifically the investigators anticipate that the CHESS effect on caregivers will be mediated by the CHESS effect on interaction patterns with clinicians, satisfaction with clinical visits and by the CHESS effect on four patient outcomes (quality of life, negative affect, average severity of nine common late-stage cancers).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast or prostate cancer patients and their primary caregivers

Exclusion Criteria:

* Cannot be homeless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2004-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Improve caregiver burden | every 2 months
Improve affect, coping, self-efficacy and information competence | every 2 months

SECONDARY OUTCOMES:
Mechanisms of CHESS effects | every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: David Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] DuBenske LL, Burke Beckjord E, Hawkins RP, Gustafson DH. Psychometric evaluation of the Health Information Orientation Scale: a brief measure for assessing health information engagement and apprehension. J Health Psychol. 2009 Sep;14(6):721-30. doi: 10.1177/1359105309338892. PMID 19687109
- [Background] DuBenske LL, Gustafson DH, Shaw BR, Cleary JF. Web-based cancer communication and decision making systems: connecting patients, caregivers, and clinicians for improved health outcomes. Med Decis Making. 2010 Nov-Dec;30(6):732-44. doi: 10.1177/0272989X10386382. Epub 2010 Nov 1. PMID 21041539
- [Result] Wen KY, Gustafson DH. Needs assessment for cancer patients and their families. Health Qual Life Outcomes. 2004 Feb 26;2:11. doi: 10.1186/1477-7525-2-11. PMID 14987334
- [Result] Dubenske LL, Chih MY, Dinauer S, Gustafson DH, Cleary JF. Development and implementation of a clinician reporting system for advanced stage cancer: initial lessons learned. J Am Med Inform Assoc. 2008 Sep-Oct;15(5):679-86. doi: 10.1197/jamia.M2532. Epub 2008 Jun 25. PMID 18579837
- [Result] DuBenske LL, Chih MY, Gustafson DH, Dinauer S, Cleary JF. Caregivers' participation in the oncology clinic visit mediates the relationship between their information competence and their need fulfillment and clinic visit satisfaction. Patient Educ Couns. 2010 Dec;81 Suppl:S94-9. doi: 10.1016/j.pec.2010.08.022. Epub 2010 Sep 28. PMID 20880656
- [Derived] Gustafson DH, DuBenske LL, Atwood AK, Chih MY, Johnson RA, McTavish F, Quanbeck A, Brown RL, Cleary JF, Shah D. Reducing Symptom Distress in Patients With Advanced Cancer Using an e-Alert System for Caregivers: Pooled Analysis of Two Randomized Clinical Trials. J Med Internet Res. 2017 Nov 14;19(11):e354. doi: 10.2196/jmir.7466. PMID 29138131
- [Derived] Chih MY, DuBenske LL, Hawkins RP, Brown RL, Dinauer SK, Cleary JF, Gustafson DH. Communicating advanced cancer patients' symptoms via the Internet: a pooled analysis of two randomized trials examining caregiver preparedness, physical burden, and negative mood. Palliat Med. 2013 Jun;27(6):533-43. doi: 10.1177/0269216312457213. Epub 2012 Sep 17. PMID 22988042